CLINICAL TRIAL: NCT05648994
Title: A Single-arm, Open-label, Dose-finding Clinical Study of TCR-T Cells in Patients With HLA-A2-expressing and NY-ESO-1-positive Recurrent or Metastatic Solid Tumors
Brief Title: TCR-T Cells for the Treatment NY-ESO-1-positive Advanced Solid Tumors
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FJ002
Record Dates: First submitted 2022-10-26; First posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-10

CONDITIONS: Solid Tumors
MeSH Terms: interventions — fludarabine; Cyclophosphamide; Albumin-Bound Paclitaxel; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TCR-T cells (Experimental): TCR-T cells will be infused to patients with advanced solid tumors after non-myeloablative lymphocyte-depleting preparative regimen.
  Interventions: Biological: TCR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide Capsules; Drug: Albumin-bound paclitaxel; Drug: IL-2

INTERVENTIONS:
Biological: TCR-T cells — patients will be administration of TCR-T cells
Drug: Fludarabine — Part of the non-myeloablative lymphocyte-depleting preparative regime
Drug: Cyclophosphamide Capsules — Part of the non-myeloablative lymphocyte-depleting preparative regime
Drug: Albumin-bound paclitaxel — Part of the non-myeloablative lymphocyte-depleting preparative regime
Drug: IL-2 — Following cell infusion, the patient will be administration high-dose IL-2.

SUMMARY:
New York Esophageal Squamous Cell Carcinoma 1 (NY-ESO-1) is a Cancer-Testis Antigen (CTA) which is expressed in various tumors. After selected the high affinity TCR gene to NY-ESO-1, the researchers insert genes into the cell that expressing a kind of protein that targeting NY-ESO-1. Then the engineered cells are re-infused in the patients with tumors for curing the tumor patient or prolonging life.

DETAILED DESCRIPTION:
This is a single-center, open-label, Phase I clinical study of TCR-T cells for the treatment of the recurrent/metastatic solid tumors patients who had failed standard therapy.

TCR-T cells are expanded from peripheral blood, and after ex vivo modification, and extensive expansion, are reinfused to patients after non-myeloablative lymphocyte-depleting preparative regimen.

The primary purpose of this study is to evaluate the safety and tolerability of TCR-T cells in patients with recurrent/metastatic solid tumors.

The second purpose of this study is to preliminarily explore the effectiveness of TCR-T cells in patients with recurrent/metastatic solid tumors.

Eligibility:

Adults aging 18-70 who were failed to standard treatment or have no standard treatment with recurrent/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Have the willingness to communicate with investigator, be able to understand and follow the trail requirements, and voluntarily to participate in the trail;
2. 18 ~70 years old (gender is not limited;)
3. The expected survival period is at least 3 months;
4. ECOG score of 0-1;
5. Patients with recurrent or metastatic solid tumors confirmed by histopathology;
6. Subjects who failed standard treatment in the past or have no standard treatment currently tor who are judged by the investigator to be unsuitable for current standard treatment for other reasons, and the objective imaging assessment is disease progression;
7. According to RECIST 1.1 standard, there is at least one measurable target lesion for efficacy evaluation;
8. NY-ESO-1 positive;
9. HLA type is HLA-A2 (except HLA-A*0203);

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding, or have a positive blood pregnancy test at baseline;
2. Subjects who have had severe allergic reactions to any drug or its components in this trial in the past;
3. Subjects who have received any investigational drug within 28 days before the infusion of TIL cells, or participated in another clinical study at the same time;
4. Subjects who have other known history of malignant tumors in the past 5 years, except for localized tumors that have been cured, including in situ cervical carcinoma, basal cell carcinoma of the skin, and in situ prostate carcinoma;
5. Patients who have received adoptive cell therapy in the past;
6. According to the judgment of the investigator, the condition of the subject is not suitable for this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity | up to Day28
  Dose Limiting Toxicity (DLT) is defined as patients with the adverse event (AE) or laboratory abnormality recognized by Investigators, and should be possibly related to TCR-T cells therapy
Adverse Event | up to 24 months
  The severity and incidence of various adverse events and serious adverse events

SECONDARY OUTCOMES:
Overall response rate (ORR) | up to 24 months
  Objective response rate (ORR) is defined as the proportion of patients in whom a complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors [RECIST 1.1]) is observed as best overall response
Progression free survival (PFS) | up to 24 months
  PFS is defined as time from start of treatment to the first documentation of disease progression or death, whichever occurs first
Overall survival | up to 24 months
  OS defined as the time from start of treatment to the date of death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong He, Principal Investigator — Fujian Cancer Hospital

IPD SHARING:
Plan to Share IPD: No